CLINICAL TRIAL: NCT01585584
Title: Triple-Therapy With PegInterferon α-2b + Ribavirin + Boceprevir in Patients With HCV Genotype 3 Who Previously Failed Treatment With PegInterferon α + Ribavirin
Brief Title: Triple-Therapy in Patients With HCV Genotype 3 Who Previously Failed Treatment
Acronym: LeeG3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Sam Lee, Hepatologist, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MISP #39897; 24411 (Other: University of Calgary)
Record Dates: First submitted 2012-04-18; First posted 2012-04-26 (Estimated); Results first posted 2015-09-21 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-08

CONDITIONS: Hepatitis C
Keywords: Boceprevir; Hepatitis C Genotype 3
MeSH Terms: conditions — Hepatitis C | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; Protease Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Boceprevir (Experimental)
  Interventions: Drug: Boceprevir

INTERVENTIONS:
Drug: Boceprevir — All patients will receive a 4-week lead-in with Peginterferon and Ribavirin therapy, followed by 24 weeks of Pegetron 1.5microg/kg + weight-based ribavirin + boceprevir 800mg tid. HCV RNA (Cobas TaqMan) will be measured at baseline and at treatment weeks 4, 6,8,12,16,20,24 and 28, and post-treatment weeks 12 and 24 (to obtain SVR-12 and SVR-24 results).
  Other Names: VICTRELIS™; boceprevir capsules, 200 mg; Hepatitis C Virus (HCV) Protease Inhibitor

SUMMARY:
The purpose of this study is to test the potential antiviral efficacy of triple-combination therapy with Peginterferon α-2b + ribavirin + boceprevir (PRB) in patients with HCV genotype 3 who previously failed Peginterferon α + ribavirin (non-responders or relapsers).

DETAILED DESCRIPTION:
i) Obtain preliminary information on the association between important baseline and on-treatment factors and SVR in this patient population. Variables to be examined may include gender, age, advanced fibrosis or cirrhosis (F3 or F4 estimated by Fibroscan), baseline viral load, RVR, wk 8 viral load, end-of-treatment viral response.

ii) Evaluate adverse events. iii) Evaluate viral resistance.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible for the study if they meet the following inclusion criteria:

  1. 18 years of age or older
  2. Infected with HCV genotype 3 (mixed genotypes are NOT permitted)
  3. Have received at least 12 weeks of previous treatment with peginterferon-α + ribavirin
  4. Detectable serum HCV-RNA
  5. No significant co-morbid conditions
  6. Liver biopsy is not necessary
  7. Cirrhotic patients will be eligible to participate if Child-Pugh class A (maximum 15% of subjects)

Exclusion Criteria:

* Subjects will be excluded from participation in this study if the following conditions are present:

  1. Significant comorbidities: uncontrolled psychiatric conditions including severe depression, cardiovascular, respiratory, renal or metabolic conditions, active carcinoma.
  2. Active substance abuse within the past 12 months
  3. Co-infection with hepatitis B or HIV
  4. Decompensated cirrhosis (Child-Pugh class B or C)
  5. Significant cytopenia - any of the following: platelets <80 x 109/L, neutropenia <1.2 x 103/L, Hb <120 g/l for men or 110 g/l for women
  6. Lack of informed consent
  7. Previous null-responders (<2 log10 decrease at week 12 with previous PR therapy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Lee, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary Liver Unit, Calgary, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was hoped that 21 patients with chronic HCV genotype 3 who had failed to achieve an SVR with a standard course of treatment with Peginterferon α + ribavirin (PR) would be selected from the University of Calgary Liver Unit (UCLU) database. 11 patients were able to be enrolled in the study.The last patient completed the study in December 2014.
Pre-assignment Details: Of the 11 patients who were enrolled in the study, 1 patient was a screen failure.
Groups:
- Victrelis Triple: All patients will receive a 4-week lead-in with peginterferon and ribavirin therapy, followed by 24 weeks of Pegetron 1.5mg/kg + weight-based ribavirin + boceprevir 800mg tid (Victrelis Triple)
Period: Overall Study
Arm/Group | Victrelis Triple
Started | 10
Completed | 6
Not Completed | 4
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Victrelis Triple
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (6.945)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Number; unit: participants]
  Canada | 10

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response (SVR) at 24 Weeks Post Treatment
Description: Sustained Virologic Response (SVR) is evaluated 24 weeks after end of treatment and defined as undetectable plasma HCV-RNA at follow up week 24. HCV RNA is measured using Cobas TaqMan.Of the 6 subjects who completed the treatment, 3 obtained SVR at 24 weeks post treatment.
Time Frame: 24 weeks after treatment
Population: Patients who completed full course of treatment
Measure: Number; unit: participants
Arm/Group | Victrelis Triple
Number analyzed (Participants) | 6
participants
  Subjects who completed treatment | 6
  Subjects who obtained SVR 24 | 3

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Victrelis Triple
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Victrelis Triple (N=10)
Emergency room visit due to suspected celulitis (Infections and infestations) | 1 (1)
Pregnancy in spouse (Reproductive system and breast disorders) | 1 (1) — Subject was instructed to use 2 methods of birth control for duration of study. however subject's partner had an unplanned pregnancy shortly after discontinuing study drug. Subject's spouse chose to terminate the pregnancy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Victrelis Triple (N=10)
Abdominal pain (General disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3
Anemia (Blood and lymphatic system disorders) | 9
Anisocytosis (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 6
Anxiety (Psychiatric disorders) | 1
Apthous ulcers (Skin and subcutaneous tissue disorders) | 2
Blurred vision (Eye disorders) | 3
Brittle nails (Skin and subcutaneous tissue disorders) | 1
Cellulitis (Infections and infestations) | 1
Chest pain (Musculoskeletal and connective tissue disorders) | 2
Chills (General disorders) | 8
Chest pain on inspiration (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Delayed healing (Blood and lymphatic system disorders) | 3
Despressed mood (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Difficulty concentrating (Psychiatric disorders) | 2
Diuresis (Renal and urinary disorders) | 3
Dizziness (Ear and labyrinth disorders) | 5
Dry mouth (General disorders) | 6
Dry nose (General disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 6
Dysgeusia (Gastrointestinal disorders) | 8
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Exerional dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Fatigue (General disorders) | 8
Feeling overwhlemed (Psychiatric disorders) | 1
Fever (General disorders) | 7
Headache (General disorders) | 7
Increased LDL (Blood and lymphatic system disorders) | 1
Hyperactivity (General disorders) | 1
Hypercholesterolemia (Blood and lymphatic system disorders) | 2
Hypertriglyceridemia (Blood and lymphatic system disorders) | 5
Hypoalbuminema (Blood and lymphatic system disorders) | 4
Hypochloremia (Blood and lymphatic system disorders) | 3
Hypochromia (Blood and lymphatic system disorders) | 1
Hyponatremia (Blood and lymphatic system disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Increased INR (Blood and lymphatic system disorders) | 3
Increased leukocytes (Blood and lymphatic system disorders) | 1
Increased neutrophils (Blood and lymphatic system disorders) | 1
Local injection site reactions (Skin and subcutaneous tissue disorders) | 9
Insomnia (General disorders) | 10
Irritability (Psychiatric disorders) | 4
Itchiness (Skin and subcutaneous tissue disorders) | 7
Joint pain (Musculoskeletal and connective tissue disorders) | 6
Leukopenia (Blood and lymphatic system disorders) | 8
Low HDL (Blood and lymphatic system disorders) | 1
Lung congestion (Respiratory, thoracic and mediastinal disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 3
Memory impairment (Psychiatric disorders) | 1
Muscle pain (Musculoskeletal and connective tissue disorders) | 9
Nausea (Gastrointestinal disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 8
Non-productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Nose bleed (Blood and lymphatic system disorders) | 3
Numbness/tingling (Nervous system disorders) | 2
Orthostatic hypotension (Cardiac disorders) | 2
Polychromasia (Blood and lymphatic system disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Worsening of psoriasis (Immune system disorders) | 2
Pulsatile tinnitus (Ear and labyrinth disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 6
Resltess legs (Nervous system disorders) | 1
Sinus congestion (General disorders) | 3
Skin tags (Skin and subcutaneous tissue disorders) | 1
Irritated eyes (Eye disorders) | 4
Peripheral edema (General disorders) | 1
Tender gums (Skin and subcutaneous tissue disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Tongue discolouration (Gastrointestinal disorders) | 1
Transient heart rate increase (Cardiac disorders) | 1
Indigestion (Gastrointestinal disorders) | 5
Vasculitis (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Weakness (Musculoskeletal and connective tissue disorders) | 2
Weight loss (General disorders) | 5
Low LDL (Blood and lymphatic system disorders) | 1

LIMITATIONS AND CAVEATS:
Small sample size (n=11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No